CLINICAL TRIAL: NCT03993626
Title: A Phase Ib/ II Trial to Assess the Safety and Efficacy of CXD101 in Combination With the PD-1 Inhibitor Nivolumab in Patients With Metastatic, Previously-Treated, Microsatellite-Stable Colorectal Carcinoma
Brief Title: A Trial of CXD101 in Combination With Nivolumab in Patients With Metastatic Microsatellite-Stable Colorectal Cancer
Acronym: CAROSELL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Celleron Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTL-101-023; 2017-004509-42 (EudraCT Number)
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Colorectal Neoplasms Malignant
MeSH Terms: conditions — Colonic Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Open label, single arm, phase 1b/2 safety; and efficacy using Simon Two-Stage analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CXD101 and Nivolumab combination (Experimental): * CXD101 will be presented as 10mg HPMC capsules and will be taken orally for 5 consecutive days repeated every three weeks on an outpatient basis.
  * Nivolumab will be presented as a 10 mg/mL solution in a single-dose vial, administered as iv infusion over 60 mins, repeated every two weeks.
  * CXD101 in combination with nivolumab will be administered in the Phase II component of the trial at doses determined in the Phase Ib component.
  Interventions: Drug: CXD101 in Combination With Nivolumab

INTERVENTIONS:
Drug: CXD101 in Combination With Nivolumab — HDAC inhibitor in combination with anti-PD-1 monoclonal antibody

SUMMARY:
This is a study to assess the safety and efficacy of CXD101 in combination with the PD-1 Inhibitor Nivolumab in patients with metastatic, previously-treated, Microsatellite-Stable (MSS) Colorectal Carcinoma (CRC). The primary hypothesis of this study is that CXD101 and anti-PD1 monoclonal antibody synergise the anti-tumour activity in MSS colorectal cancer patients (~95% of CRC) who do not seem to respond to anti-PD1 or -PD-L1 immunotherapy alone.

DETAILED DESCRIPTION:
Phase Ib trial: This single-arm dose escalation trial will determine the safety, tolerability and dose limiting toxicities (DLT) and therefore the maximum tolerated dose (MTD) of repeat doses of nivolumab combined with CXD101. The incidence and severity of adverse events (evaluated according to CTCAE version 4.03), vital signs, ECG parameters, biochemistry, haematology and urinalysis will be recorded to determine tolerability.

Dose escalation will proceed as follows:

Dose Level 1 Nivolumab 240 mg iv q 2 weekly; with CXD101 30 mg (20mg mane, 10mg nocte) po for 5 days q 3 weekly (n=3-6) with both drugs commencing on the same day in cycle 1.

Dose Level 2 Nivolumab 240 mg iv q 2 weekly; with CXD101 40mg (20 mg bid) po for 5 days q 3 weekly (n=6) with both drugs commencing on the same day in cycle 1.

A maximum of 15 subjects will be required.

Phase II trial: Following completion of the Phase Ib study, a Phase II CXD101/ nivolumab combination dose will be selected by the Data and Safety Monitoring Committee. Up to a further 40 subjects will then be treated at the selected Phase II CXD101/ nivolumab combination dose. Subjects may continue to receive CXD101/ nivolumab until complete response, disease progression, unacceptable toxicity, withdrawal of consent, or other medical problems supervene.

Efficacy will be measured using Immune Response Evaluation Criteria in Solid Tumours (iRECIST) Imaging studies, typically CT scan of chest, abdomen & pelvis, supplemented by MRI of liver when required, will be performed at Baseline and after every 6 weeks, with objective confirmation of response 6 weeks (+/- 1 week) after observation. Safety parameters will be assessed as in the Phase I study. In addition there will be a series of translational analyses including correlation of tumour biomarker expression with response.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Biopsy-confirmed MSS, MMR-P CRC. It is acceptable for this test to be performed on the archived primary colorectal cancer tissue and repeat biopsy for MSS testing is not required unless assay not yet performed and insufficient material available
* Previous first and second line treatment (unless contra-indicated) including use of oxaliplatin and irinotecan unless documented intolerance of these
* Measurable disease: longest diameter≥10mm (short axis ≥15mm for nodal lesions)
* Age > 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Predicted life expectancy > 3 months
* Adequate organ and bone marrow function: Hb> 10.0g/dL (may be transfused to this level), neutrophils> 1.5x10^9/L and platelets> 100x10^9/L
* Female patients with reproductive potential must have a negative urine and serum pregnancy test prior to starting treatment. Both women of reproductive potential and men must agree to use a medically acceptable method of contraception throughout the treatment period and for 5 months after discontinuation of treatment (i.e., combined oestrogen and progestogen ovulation inhibition; progestogen-only ovulation inhibition; intrauterine device; intrauterine hormone-releasing system; bilateral tubal occlusion; or vasectomised partner). Oral contraception and parenteral hormonal contraceptives (patches, injectables and implants) that may be affected by enzyme-inducing drugs should only be used in combination with a barrier method. All males with partners of childbearing potential or whose partners are pregnant must use barrier contraception for the duration of dosing and for 5 months post-dosing.

Exclusion Criteria:

* Pregnant or breast feeding
* Pre-existing auto-immune conditions
* Medical conditions requiring systemic immunosuppression
* Previous treatment with an HDAC inhibitor or PD-1/PD-L1 inhibitor
* Other chemotherapy, radiotherapy, or investigational therapy within 4 weeks of the Screening /Baseline Assessment
* Unresolved clinically significant toxicity from a previous treatment
* History of recent active chronic inflammatory bowel disease and/or bowel obstruction
* Renal function: Serum creatinine > 1.5 x ULN, or creatinine clearance < 60mL/min (Cockcroft-Gault formula)
* Liver function: AST > 3.0 x ULN; OR total bilirubin > 1.5 x ULN
* Clinically significant myocardial infarction, severe/unstable angina pectoris, congestive heart failure NYHA Class III or IV, or pulmonary disease within 6 months
* Symptomatic brain metastasis, uncontrolled seizure disorder, spinal cord compression, or carcinomatous meningitis
* Clinically significant active infection requiring antibiotic or antiretroviral therapy
* History of malignancy other than MSS CRC, unless there is the expectation that the malignancy has been cured, and tumour specific treatment for the malignancy has not been administered within the previous 5 years
* History of pneumonitis, immune hepatitis or myocarditis, or current uncontrolled thyroid disease
* Current positive serology for Hepatitis B or C virus
* History of any allergy to excipients of the Investigational Medicinal Products (sodium citrate dihydrate, sodium chloride, mannitol, pentetic acid, Polysorbate 80, sodium hydroxide, hydrochloric acid, hydroxypropyl methylcellulose)
* Receipt of any live vaccine 30 days or fewer prior to administration of first dose IMP
* Inability to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2019-12-15 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Immune Disease Control Rate (iDCR) | 6 months
  complete response [iCR], partial response [iPR], and stable disease [iSD] rate) after Seymour et al, 2017.

SECONDARY OUTCOMES:
20-week immune-related progression-free survival (PFS) | 20 weeks
  Progression-free survival will be measured from the date of first dose until death from any cause, with measurement cut-off at 20 weeks. Subjects who discontinue from treatment will classed as "censored" at the last timepoint when their PFS status was known. Subjects who discontinue from the study will be classed as "censored" at the time they discontinue.
  A Kaplan-Meier survival curve will be plotted and the 20-week PFS rate determined, with a 95% confidence interval.
Best Objective Response Rate | 6 months
  iCR + iPR / iCR + iPR + iSD + iPD x 100. The Objective Response Rate will be calculated as the combined percentage of subjects who have achieved as best response: complete response, or partial response.
Overall Survival (OS) | 6 months
  Overall Survival will be measured from the date of first dose until death from any cause. Subjects who discontinue from treatment will be followed up for survival but will be classed as "censored" at the last timepoint when their survival status was known. Subjects who discontinue from the study will be classed as "censored" at the time they discontinue.
  A Kaplan-Meier survival curve will be plotted for overall survival.
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | 6 months
  AEs may be directly observed, evident in laboratory or diagnostic results, reported spontaneously by the subject, or by questioning the subject at each study visit. All subjects who complete screening, receive at least one dose of study medication and who have at least one safety assessment (including "death") will be in the Safety Set.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Kerr, MD, Principal Investigator — Department of Oncology, University of Oxford
Locations (1):
- Celleron Therapeutics Ltd, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No